CLINICAL TRIAL: NCT01164670
Title: Evaluation of the Reproducibility of Jumping Mechanography in Older Adults and Comparison With Current Functional Assessment Tools
Brief Title: Evaluation of the Reproducibility of Jumping Mechanography
Acronym: Jump
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: H-2010-0011
Record Dates: First submitted 2010-07-15; First posted 2010-07-19 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2011-03

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum will be collected for measurement of laboratory studies (serum chemistries, TSH and 25[OH]D),
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Men: Men over 70 years old.
- Women: Women over 70 years old.

SUMMARY:
Sarcopenia, the age-related decline in muscle mass and function (widely recognized as "frailty"), is increasingly being appreciated, primarily in the research environment. Interventions to prevent or treat sarcopenia can be anticipated to reduce falls, fractures and thereby to facilitate independence and improve quality of life for older adults. Unfortunately, there is no current consensus definition of sarcopenia, thereby impeding clinical recognition and treatment. It has been advocated that low appendicular (arm and leg) lean mass, as measured by DXA, be utilized as a clinical diagnostic tool to define sarcopenia. While such an approach is possible, however, muscle strength loss is more rapid than mass loss, indicating deterioration of muscle "quality." Muscle quality may be affected by changes at the neuromuscular, cellular or subcellular levels; parameters not detected by measuring mass alone. Clearly, tools evaluating muscle performance, not simply mass, are needed to optimally identify, and subsequently monitor, treatment of older adults with sarcopenia. While current tests of muscle power/function (e.g., chair-rising, self-selected gait velocity, etc.) do correlate with functional limitation in older adults, these existing tests have limitations in that they cannot be performed in all people, may have "yes/no" results rather than a continuous scale and may not be highly precise. Thus, improved muscle function assessment tools are needed, both clinically and in research venues. Jumping mechanography is very likely one such methodology.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory, community dwelling men and women age ≥ 70 years
* Able and willing to sign informed consent
* Able to stand without assistance

Exclusion Criteria:

* Abnormalities on screening laboratory assessment deemed to be clinically significant by the study investigators
* History of myocardial infarction within the prior six months or ongoing angina
* History of injury or surgery within the prior six months which limits the ability to ambulate
* History of severe end-organ disease, e.g., cardiovascular, hepatic, hematologic, pulmonary, etc., which might limit the ability to complete this study
* History of malignancy with metastasis to the musculoskeletal system
* Neuromuscular disease impairing balance to the degree of not being able to stand without assistance
* BMD T-score of less than -3.5 at any measured site and a prior hip or vertebral fracture

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Ambulatory community dwelling adults who are able to stand without assistance. Both men and women age ≥ 70 years from the Madison Wisconsin area. Specifically, participants will be enrolled using the following strata in each gender group: low vitamin D/low functional status (12 men and 12 women), normal vitamin D/low functional status (12 men and 12 women), low vitamin D/high functional status (12 men and 12 women), and normal vitamin D/high functional status (12 men and 12 women). Low vitamin D will be defined as 25(OH)D concentrations < 25 ng/ml, normal vitamin D status will be defined as 25(OH)D concentration of 30 ng/ml or greater. Functional status will be based on screening short physical performance battery (SPPB) score dichotomized at <9 vs. 9 and above.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2010-05; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Binkley, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Osteoporosis Clinical Center and Research Program, Madison, Wisconsin, United States